CLINICAL TRIAL: NCT02041260
Title: A Phase II Trial of Cabozantinib for the Treatment of Radioiodine (RAI)-Refractory Differentiated Thyroid Carcinoma (DTC) in the First-line Setting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 28313
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Differentiated Thyroid Cancer (DTC); Poorly Differentiated Thyroid Cancer
Keywords: Adult; differentiated thyroid cancer (DTC),; poorly differentiated thyroid cancer; not anaplastic thyroid cancer
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label Cabozantimib (Experimental)
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib

SUMMARY:
Phase II, non-randomized, open-label study to determine the efficacy of cabozantinib as a firstline treatment for patients with differentiated thyroid cancer (DTC). Subjects will receive drug at a starting dose of 60mg PO QD. Subjects can receive drug as long as they continue to derive clinical benefit or until they experience unacceptable drug-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologic or cytologic diagnosis of a DTC tumor (including poorly differentiated thyroid cancer but not anaplastic thyroid cancer) that is metastatic or unresectable and fulfills the following criteria: a. Subjects must have progressive disease as defined by RECIST 1.1 criteria when comparing baseline scans to those obtained within the prior 14 months AND b. Subject must have RAIrefractory disease based on at least one of the following: i. Prior dose of RAI exceeding 600mCi ii.Progression of disease within 18 months following a dose of 100mCi iii. Presence of target lesions as defined by modified RECIST criteria which do not take up RAI.
* The subject has had an assessment of all known disease sites eg, by computerized tomography (CT) scan, magnetic resonance imaging (MRI), bone scan as appropriate, within 28 days before the first dose of cabozantinib
* The subject is 18 years old on the day of consent.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The subject has organ and marrow function and laboratory values as follows within 4 days prior to the first dose of cabozantinib: a. Absolute neutrophil count (ANC) 1500/mm3without colony stimulating factor support b. Platelets 100,000/mm3 c. Hemoglobin 9 g/dL d.Bilirubin 1.5 the upper limit of normal (ULN). For subjects with known Gilberts disease, bilirubin 3.0mg/dL e. Serum albumin 2.0 g/dl f. Serum creatinine 1.5 ULN or creatinine clearance (CrCl) 50 mL/Page 9 of 16 min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used: Male: CrCl(mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72) Female: Multiply above result by 0.85 g.Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 3.0 ULN h. Lipase 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis i. Urine protein/creatinine ratio (UPCR) 1 j. Serum phosphorus, calcium, magnesium and potassium LLN
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).
* Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as amenorrhea 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason.
* An archived tumor specimen is available for collection.

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy),biologic agents (eg, cytokines or antibodies), or any other anti-cancer systemic therapy (including multi-kinase inhibitors).
* Prior treatment with cabozantinib
* The subject has received radiation therapy: a. to the thoracic cavity, abdomen or pelvis within 3 months of the first dose of study treatment thathas with ongoing complications or is without complete recovery and healing (CT changes related to radiation treatment which are not clinical significant are allowed). b. to bone or brain metastasis within 14 days of the first dose of study treatment c. to any other site(s) within 28 days of the first dose of study treatment
* The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* The subject has not recovered to baseline or CTCAE Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs (eg. albumin).
* The subject has a primary brain tumor.
* The subject has active brain metastases or epidural disease who have not been treated with radiation therapy (Note: Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 2 months before starting study treatment. (Baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility.)
* The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test 1.3 the laboratory ULN within 7 days before the first dose of study treatment.
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin ( 81 mg/day), low-dose warfarin (1mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted.
* The subject requires chronic concomitant treatment of strong CYP3A4 inducers (eg, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. Johns Wort).
* The subject has experienced any of the following: a. clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment b. hemoptysis of 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment c. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor in contact with, invading or encasing any major blood vessels
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions: a. Cardiovascular disorders including i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening ii. Concurrent uncontrolled hypertension defined as sustained BP 140 mm Hg systolic, or 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment iii. Any history of congenital long QT syndrome iv.

Any of the following within 6 months before the first dose of study treatment: unstable angina pectoris clinically-significant cardiac arrhythmias stroke (including TIA, or other ischemic event) myocardial infarction thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study) b. Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including: i. Any of the following within 28 days before the first dose of study treatment intra-abdominal tumor/metastases invading GI mucosa active peptic ulcer disease, inflammatory bowel disease (including ulcerative colitis and Crohns disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis malabsorption syndrome ii. Any of the following within 6 months before the first dose of study treatment: abdominal fistula gastrointestinal perforation bowel obstruction or gastric outlet obstruction intra-abdominal abscess.Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months before the first dose of study treatment. c. Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy d. Other clinically significant disorders such as: i. active infection requiring systemic treatment within 28 days before the first dose of study treatment ii. serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment iii. history of organ transplant iv. concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment v. history of major surgery as follows: (1) Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications (2) Minor surgery within 1 months of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications In addition complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery

* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) 500 ms within 28 days before randomization. . Note: if initial QTcF is found to be 500 ms, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is 500 ms, the subject meets eligibility in this regard
* The subject is pregnant or breastfeeding.
* The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation. 21. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Brose, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not at this time